CLINICAL TRIAL: NCT03027323
Title: Washington Study of AxoTrack-Guided Central Venous Cannulation
Acronym: WASHCAN
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study not funded; no participants enrolled
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Graham Nichol, Professor, School of Medicine: General Internal Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00000958
Record Dates: First submitted 2017-01-19; First posted 2017-01-23 (Estimated); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Hypotension
Keywords: undifferentiated hypotension; central venous cannulation
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- AxoTrack System guided CVC insertion (Other): AxoTrack System guided CVC
  Interventions: Device: AxoTrack System
- CVC insertion guided by landmark (No Intervention): Anatomical landmarks to guide CVC

INTERVENTIONS:
Device: AxoTrack System — The AxoTrack system is a novel ultrasound guidance system intended to facilitate central venous cannulation (CVC) by a single operator as well as to reduce complications and time associated with CVC. The AxoTrack has a small ultrasound scan head which facilitates imaging of the subclavian vein.
  Arms: AxoTrack System guided CVC insertion

SUMMARY:
Undifferentiated hypotension is a medical emergency where a patient's blood pressure drops to critical levels due to several possible reasons. The medical staff treating the patient will need to find out the reason for your drop in blood pressure as soon as possible. When treating low blood pressure, the medical staff typically performs a procedure called central venous cannulation (CVC). CVC involves accessing a large vein (usually the subclavian under the collarbone) by inserting a needle into the vein. By doing this, the medical staff can measure the pressures in the patient's veins or give medicine to the patient while they are in the hospital.

The purpose of this study is to compare the time needed to complete CVC using the AxoTrack device to CVC guided by landmarks on a patient's body. The investigators expect that there will be a maximum of 30 patients enrolled in this study.

DETAILED DESCRIPTION:
Central venous cannulation (CVC) is commonly performed to give volume resuscitation and parenteral medications to patients with time sensitive conditions such as severe traumatic injury or undifferentiated shock. CVC via the subclavian route is associated with more frequent technical complications but less frequent infection or thrombosis as compared with via the internal jugular or femoral veins. Traditionally CVC via the subclavian vein is guided by anatomical landmarks. CVC guided by real-time use of traditional diagnostic ultrasound device is associated with a lower technical failure rate (overall and on first attempt), fewer punctures, faster access, and fewer mechanical complications as compared with guidance by anatomical landmarks when performed via the internal jugular vein. It remains unclear whether CVC guided by real-time ultrasound is associated with significantly lower failure and complication rates as compared with CVC guided by landmarks when performed via the subclavian vein. CVC guided by real-time ultrasound may reduce the incidence of complications, number of punctures, and the time between skin penetration and the aspiration of venous blood into the syringe as compared with guidance by landmarks. A limitation of guidance by a traditional diagnostic ultrasound device is it that it may require an assistant to perform, which may not be feasible when treating time sensitive conditions or in low resource settings. In addition, most traditional ultrasound probes are not designed to image the subclavian vein behind the clavicle. The AxoTrack system is a novel ultrasound guidance system recently cleared for human use by the United States Food and Drug Administration. It is intended to facilitate CVC by a single operator as well as to reduce complications and time associated with CVC. The AxoTrack has a small ultrasound scan head which facilitates imaging of the subclavian vein. It remains unclear whether CVC guided by AxoTrack reduces procedure times and complication rates when compared with CVC using landmark guidance in patients with undifferentiated hypotension.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed systolic blood pressure < 90 mmHg in emergency department;
2. Aged at least 18 years; and
3. Need for CVC in emergency department.

Exclusion Criteria:

1. Preexisting written do not attempt resuscitation order;
2. Prisoners;
3. Pregnant;
4. ST-elevation on initial 12-lead electrocardiogram;
5. Blunt or penetrating traumatic injury;
6. Major burn;
7. Exsanguination;
8. Obese (i.e. estimated body mass index > 30 kg/m2);
9. Known coagulation disorders;
10. Contraindication to CVC by subclavian route; or
11. Patients in extremis for whom placement of the device would delay emergent care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-02-10 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Time to insertion of CVC into a subclavian vein | 0-30 minutes
  The time it takes for the care provider to insert the central venous cannulation device into the subclavian vein

CONTACTS AND LOCATIONS:
Overall Officials: Graham Nichol, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No